CLINICAL TRIAL: NCT06978374
Title: Ultrasonographic Evaluation of Thoracolumbar Fascia Morphology in Axial Spondyloarthropathy and Controls: A Pilot Study With Clinical Assessment of Myofascial Trigger Points
Brief Title: Ultrasonographic Assessment of Thoracolumbar Fascia in AxSpA and Controls With Trigger Point Evaluation
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Yuzlem Gyuner SIDZHIMLI MD, Principal Investigator, Ankara University
Other Study IDs: AUPMRYGSThesis
Record Dates: First submitted 2025-05-03; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Axial Spondylarthritis (axSpA); Myofascial Trigger Point Pain (MTrP); Ultrasound Exams
Keywords: Thoracolumbar fascia; Axial Spondyloarthropatis (axSpA); Myofascial Trigger Point Pain (MTrP); Ultrasound; Sonography
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- AxSpA group: This study included individuals aged between 18 and 65 years who were classified as having axial spondyloarthritis (axSpA), including both radiographic and non-radiographic forms, according to the Assessment of SpondyloArthritis International Society (ASAS) classification criteria. Participants with additional health conditions that could affect thoracolumbar fascia (TLF) morphology or spinal biomechanics were excluded from the study. Exclusion criteria included: History of severe back or lower extremity trauma or surgery, Significant spinal deformity (e.g., scoliosis, kyphosis, spinal stenosis), History of spinal surgery, History of spinal fracture, Malignancy or spinal infection, Neurological deficit due to nerve root compression, Neurological or major psychiatric disorders, Bleeding disorders, Previous lumbar steroid injection or current systemic steroid use, Pregnancy, Disability status or ongoing legal process related to low back pain, Presence of acute systemic infection
  Interventions: Other: Sonographic examination of thoracolumbar fascia, manual examination of MTrP
- Healthy group: Participants in the healthy control group were age-matched (18-65 years) and selected according to the same exclusion criteria applied to the patient group.
  Interventions: Other: Sonographic examination of thoracolumbar fascia, manual examination of MTrP

INTERVENTIONS:
Other: Sonographic examination of thoracolumbar fascia, manual examination of MTrP — Patients were positioned in the prone position, with a cushion placed under the abdomen to flatten the lumbar lordosis.
  A 14-18 MHz linear transducer was used for ultrasonographic (USG) evaluation, performed with a GE Logiq P5 ultrasound device (Serial No: GE-114118SU3).
  The USG probe was placed longitudinally at the L2-L3 intervertebral level, 2 cm lateral to the vertical line connecting the spinous processes on both sides, in order to assess the thoracolumbar fascia (TLF).

SUMMARY:
The goal of this observational study is to evaluate whether changes in the thoracolumbar fascia (TLF)-a connective tissue in the lower back-are related to pain and disease severity in patients with axial spondyloarthropathy (ax-SpA), a chronic inflammatory spine condition. The study involves adults diagnosed with ax-SpA and healthy volunteers of similar age and gender.

The main questions it aims to answer are:

Is the thickness or shape of the thoracolumbar fascia different in patients with ax-SpA compared to healthy individuals? Is there a relationship between changes in the thoracolumbar fascia and the presence of painful muscle trigger points? Researchers will compare measurements in ax-SpA patients and healthy volunteers to see if differences in fascia structure are linked to pain, function, and disease activity.

Participants will:

Undergo a back ultrasound (non-invasive imaging) to assess the thickness and structure of the thoracolumbar fascia.

Be examined for muscle trigger points using gentle manual palpation. Complete questionnaires and assessments on physical function, quality of life, and disease activity.

DETAILED DESCRIPTION:
The goal of this observational study is to explore whether structural changes in the thoracolumbar fascia (TLF)-a connective tissue layer in the lower back-are related to pain, stiffness, and disease activity in individuals with axial spondyloarthropathy (ax-SpA), a chronic inflammatory condition that affects the spine and can cause significant back pain and limited mobility. The study also examines whether these changes are linked to myofascial trigger points, which are sensitive or painful spots in the muscles.

This research includes adults diagnosed with ax-SpA, as well as healthy volunteers of similar age and gender who do not have chronic back pain or spinal diseases.

The main questions it aims to answer are:

Do patients with ax-SpA have increased thickness or irregular structure in the thoracolumbar fascia compared to healthy individuals? Is there a connection between fascia changes and the presence of painful muscle trigger points? Are these findings related to the severity of disease symptoms, such as pain, stiffness, physical function, and quality of life? Does the use of anti-inflammatory or immune-modulating medications affect the presence of these muscle trigger points? Researchers will compare ultrasound and clinical findings between ax-SpA patients and healthy volunteers to determine whether structural differences in the fascia can be used as a non-invasive indicator of disease burden.

Participants will:

Undergo a high-resolution ultrasound scan of their lower back to assess the structure and thickness of the thoracolumbar fascia.

Receive a manual examination to check for muscle trigger points in the lower back.

Complete questionnaires related to pain, function, fatigue, and quality of life.

Share information about their medical history, including the use of medications such as non-steroidal anti-inflammatory drugs (NSAIDs), disease-modifying antirheumatic drugs (DMARDs), and TNF-alpha inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 65 years
* Diagnosis of axial spondyloarthritis (axSpA) according to the Assessment of -SpondyloArthritis International Society (ASAS) classification criteria, or being a healthy control with no known musculoskeletal or systemic inflammatory disease
* Ability to lie in the prone position for ultrasonographic examination
* Willingness to participate in the study
* Provision of written informed consent prior to inclusion

Exclusion Criteria:

* History of significant back or lower extremity trauma or orthopedic surgery
* Presence of major spinal deformities (e.g., scoliosis, kyphosis, spinal stenosis)
* History of spinal surgery or spinal fracture
* Known malignancy or spinal infection
* Neurological deficits due to nerve root compression
* Presence of a diagnosed neurological or major psychiatric disorder
* Known bleeding disorders
* History of lumbar steroid injection or current use of systemic corticosteroids
* Current pregnancy
* Legal or disability status related to low back pain
* Presence of an acute systemic infection
* Refusal or inability to provide written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult male and female participants aged 18 to 65 years, who presented to the Rheumatology outpatient clinics of Ankara University School of Medicine Hospital, including individuals diagnosed with axial spondyloarthritis based on ASAS criteria and healthy controls who provided written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic Assessment of Thoracolumbar Fascia (TLF) Thickness | Baseline (Day 1)
  Thickness of the thoracolumbar fascia (TLF) will be measured using musculoskeletal ultrasound at the L2-L3 vertebral level, bilaterally.
  Unit of measures: millimeters (mm)
Thoracolumbar fascia morphology | Baseline (Day 1)
  The morphology of the thoracolumbar fascia will be evaluated bilaterally as either regular or irregular based on ultrasonographic appearance at the same level.
  Unit of Measure: Categorical (Regular/Irregular)
Presence of myofascial trigger points | Baseline (Day 1)
  Presence or absence of myofascial trigger points will be assessed through standardized manual palpation criteria during clinical examination.
  Unit of Measure: Binary (Present/Absent)

SECONDARY OUTCOMES:
Correlation between thoracolumbar fascia thickness and presence of myofascial trigger points | Baseline (Day 1)
  A correlation analysis will be performed between thoracolumbar fascia thickness (measured in mm via ultrasound) and the presence or absence of myofascial trigger points (determined by physical examination).
Correlation between thoracolumbar fascia morphology and presence of myofascial trigger points | Baseline (Day 1)
  A correlation will be evaluated between fascia morphology (categorized as regular/irregular on ultrasound) and the presence or absence of myofascial trigger points.

CONTACTS AND LOCATIONS:
Overall Officials: Sebnem ATAMAN, Study Chair, Study Chair — Ankara University School of Medicine, Department of Rheumathology; Yuzlem Gyuner SIDZHIMLI, MD, Principal Investigator — Ankara University School of Medicine, Department of Physical Medicine and Rehabilitation; Seçilay GÜNEŞ, Ass Prof, Study Director — Ankara University School of Medicine, Department of Physical Medicine and Rehabilitation
Locations (1):
- Ankara University, Faculty of Medicine Hospital, Ankara, Mamak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical and privacy considerations, as well as institutional policy regarding the handling of sensitive clinical data in non-interventional studies.

REFERENCES:
- [Background] De Coninck K, Hambly K, Dickinson JW, Passfield L. Measuring the morphological characteristics of thoracolumbar fascia in ultrasound images: an inter-rater reliability study. BMC Musculoskelet Disord. 2018 Jun 1;19(1):180. doi: 10.1186/s12891-018-2088-5. PMID 29859080
- [Background] Abe H, Hayashi S, Kim JH, Murakami G, Rodriguez-Vazquez JF, Jin ZW. Fetal development of the thoracolumbar fascia with special reference to the fascial connection with the transversus abdominis, latissimus dorsi, and serratus posterior inferior muscles. Surg Radiol Anat. 2021 Jun;43(6):917-928. doi: 10.1007/s00276-020-02668-4. Epub 2021 Jan 12. PMID 33438110
- [Background] Boccon Gibod L, Correas G, Godefroy D, Ducellier R, Teyssier P. [Radio-transparent renal calculi and epithelial tumours. Contribution of ultrasound and CT scan to the diagnosis (author's transl)]. Nouv Presse Med. 1981 Oct 31;10(39):3231-2. French. PMID 7301552
- [Background] Kondrup F, Gaudreault N, Venne G. The deep fascia and its role in chronic pain and pathological conditions: A review. Clin Anat. 2022 Jul;35(5):649-659. doi: 10.1002/ca.23882. Epub 2022 Apr 27. PMID 35417568
- [Background] Hodges PW, Danneels L. Changes in Structure and Function of the Back Muscles in Low Back Pain: Different Time Points, Observations, and Mechanisms. J Orthop Sports Phys Ther. 2019 Jun;49(6):464-476. doi: 10.2519/jospt.2019.8827. PMID 31151377